CLINICAL TRIAL: NCT00508885
Title: The Effect of Oral Niacinamide on Plasma Phosphorus Levels in Peritoneal Dialysis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC 06-0462
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Last update posted 2007-07-30 (Estimated); Status verified 2007-07

CONDITIONS: Hyperphosphatemia
Keywords: hyperphosphatemia; niacinamide; ESRD; peritoneal dialysis; renal osteodystrophy
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Niacinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Niacinamide starting at 250 mg twice daily titrated up to 750 mg twice daily
  Interventions: Drug: Niacinamide
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Niacinamide — Niacinamide 250 mg twice daily titrated up to 750 mg twice daily
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
Hyperphosphatemia is common in the peritoneal dialysis population. Current strategies are insufficient to optimize phosphorus control. Animal studies have shown niacinamide, a form of vitamin B, to reduce phosphate uptake by the rat small intestine. Our trial investigates the use of niacinamide, in addition to standard phosphorus lowering strategies, to reduce plasma phosphorus levels in peritoneal dialysis patients versus placebo.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled 8-week clinical trial to evaluate the efficacy of niacinamide versus placebo to reduce plasma phosphorus levels in peritoneal dialysis patients. Patients on a stable regimen of phosphate binders with plasma phosphorus levels > 4.9 mg/dL are eligible for enrollment and randomization. The study will span 8 weeks of active medication treatment. The primary end-point will be absolute change in plasma phosphorus levels. Sixteen patients (8 randomized to each treatment arm) are needed to detect a 1.5 mg/dL difference assuming a standard deviation of 1 and powered at 80% (alpha 0.05). Placebo will be packaged to resemble the study drug in all physical attributes. The starting dose of niacinamide will be 250 mg twice daily to be titrated to 500 mg twice daily at the end of week 2 with a final titration to 750 mg twice daily at the end of week 4. Secondary end-points will include absolute change in the calcium-phosphorus product, intact parathyroid hormone, hemoglobin, platelet count, total cholesterol, HDL cholesterol, and percentage change in plasma phosphorus.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Capable of giving informed consent
* Duration of peritoneal dialysis > 3 months
* Dose of phosphate binder(s) stable over previous 2 week period
* Plasma phosphours > 4.9 mg/dL based on most recent laboratory data within 1 month of enrollment

Exclusion Criteria:

* Pregnancy
* Known liver disease
* Active peptic ulcer disease
* Treatment with carbamazepine
* Intolerance to niacinamide or niacin
* Current medication regimen including niacin or niacinamide > 100 mg daily
* Planned or expected surgical procedure in the next 4 months
* Patients in nursing home or extended care facilities where administration of the study drug may not be appropriately given

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-10; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The change in plasma phosphorus after 8 weeks of niacinamide versus placebo | 8 weeks

SECONDARY OUTCOMES:
The change in intact parathyroid hormone, calcium-phosphorus product, cholesterol profile, and percentage change in plasma phosphorus | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O Young, MD, Principal Investigator — Washington University, Renal Division
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Young DO, Cheng SC, Delmez JA, Coyne DW. The effect of oral niacinamide on plasma phosphorus levels in peritoneal dialysis patients. Perit Dial Int. 2009 Sep-Oct;29(5):562-7. PMID 19776051